CLINICAL TRIAL: NCT00205764
Title: Randomised, Non-blind, Parallel Group Study to Compare Tandem High Dose Melphalan (200mg/m²) Versus Triple Intermediate Dose Melphalan (100mg/m²) and Stem Cell Transplantation in Induction Phase and Prednisolone/IFN Versus IFN in Maintenance Therapy in Newly Diagnosed Patients With Multiple Myeloma
Brief Title: Tandem High Dose Melphalan Versus Triple Intermediate Dose Melphalan and Stem Cell Transplantation in Induction Phase and Prednisolone/IFN Versus IFN in Maintenance Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Forum Against Cancer (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/99
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; first line tretment; high dose chemotherapy; stem cell transplantation; maintenance therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

INTERVENTIONS:
Drug: Melphalan

SUMMARY:
This is an international,multicenter, prospective, open, double randomised and controlled phase III study to compare the therapeutic efficacy of tandem high dose Melphalan versus triple intermediate dose Melpahaln in newly-diagnosed myeloma patients

DETAILED DESCRIPTION:
Patients will be enrolled into this protocol before start of Induction therapy which consists of 3 cycles or VAD with a 4 week interval followed by 1 cycle of IEV after which stem cell harvesting is performed. After stem cell harvesting is completed Patients will be randomised to one of the high dose therapy arms after response evaluation (Complete remission, Partial remission or stable disease). One group is receiving 2 Cycles of Melphalan 200mg/m² each followed by stem cell transplantation, the other group is receiving 3 Cycles of Melphalan 100mg/m² also followed by stem cell transplantation each time.

After completing high dose therapy patients will be randomised into Maintenance responding with CR, PR or SD. The maintenance therapy will be continued until relapse or progression of disease as defined by the response criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed multiple myeloma of either IgG, IgG, IgD, IgE, IgM (but excluding Waldenstöm´s macroglobulinemia) lambda of kappa light chain, low-secretory, non-secretory disease or plasma cell leukemia
* Performance status of 0, 1, 2, or 3
* Patients not pre-treated with cytostatic drugs
* Patients who clearly require treatment (usually Durie and Salmon stage II or III)
* Patients in stage I who are symptomatic and/or show progression of their disease
* Patients must have an anticipated life expectancy of at least 3 months
* Patients must have adequate organ function
* Patients must have had a minimum recovery period of 2 weeks following any major surgical procedure before entry into this study
* Patients must be between 19 and 70 years of age, also it is understood that most of the patients above 65 will not be eligible because of poor performance status or multimorbidity
* Women of childbearing potential must have a negative pregnancy test and must take adequate precautions to prevent pregnancy during treatment
* Patients must have signed an informed consent

Exclusion Criteria:

* Patients with more than 3 irradiation fields
* Patients presenting initially with one of the following conditions:
* Extramedullary plasmacytoma or solitary plasmacytoma
* Monoclonal gammopathy of undetermined significance
* Smouldering myeloma
* Patients with an irreversible performance status of 4
* Medical of psychiatric conditions that compromise the patient´s ability to give informed consent or complete the study
* Patients with congestive heart failure, NYHA III, IV
* Known HIV positivity
* Known intolerance to any of the study drugs or components
* Acute infection requiring systemic antibiotics at study entry until fully resolved
* Patients with any underlying medical condition which cannot be adequately controlled
* Patients with second primary malignancies (with the exception of cervical carcinoma in situ and non-melanoma skin malignancies) are not eligible unless the patient has been disease-free for at least five years

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 1999-03; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure

SECONDARY OUTCOMES:
Response rate
Time to response
Tolerance of treatment
Quality of life
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, MD,Univ.Prof, Principal Investigator — Wilhelminenspital 1st medical dep.-center for oncology and hematology
Locations (1):
- Wilhelminenspital, 1st Medical Department-center for oncology and hematology, Vienna, Austria